CLINICAL TRIAL: NCT06589531
Title: 6 Mm Shunt Transjugular Intrahepatic Portosystemic Shunt in Patients with Severe Liver Atrophy and Variceal Bleeding:A Prospective Single-center Randomized Controlled Study
Brief Title: Small Diameter TIPS in Patients with Severe Liver Atrophy and Variceal Bleeding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huang Mingsheng (Other)
Responsible Party: Sponsor-Investigator, Huang Mingsheng, Director of Interventional Radiology, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: II2024-234-02
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Portal Hypertension Related to Cirrhosis
Keywords: Portal hypertension; TIPS; shunt diameter; hepatic encephalopathy; stent patency
MeSH Terms: conditions — Hypertension, Portal; Hepatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 6-mm shunt TIPS group (Experimental): The diameter of TIPS covered stent is 6mm.
  Interventions: Device: During TIPS operation, shunt diameter or diameter of covered stent
- 8-mm shunt TIPS (Active Comparator): The diameter of TIPS covered stent is 8mm.
  Interventions: Device: During TIPS operation, shunt diameter or diameter of covered stent

INTERVENTIONS:
Device: During TIPS operation, shunt diameter or diameter of covered stent — Transjugular intrahepatic portosystemic shunt (TIPS) is an effective treatment strategy for managing portal hypertension-related variceal bleeding. However, the appropriate diameter of the covered stent during the TIPS procedure remains a subject of debate. To date, there is a lack of strong evidence regarding the most suitable covered stent diameter.
  Due to the lack of a dedicated 6-mm covered stent, we first released a 6-mm diameter stent (SD Express; Boston Scientific Co., or Luminexx; Bard Medical Division) in the liver parenchymal segment of the shunt, and then released an 8-mm TIPS stent (Viatorr; WL Gore & Associates) to create a final 6-mm shunt.
  Arms: 6-mm shunt TIPS group
Device: During TIPS operation, shunt diameter or diameter of covered stent — After successful puncture, in the 8-mm shunt group, a balloon with a diameter of 6 mm was used to expand the shunt, and then an 8-mm covered stent was implanted (Viatorr; WL Gore & Associates, Inc.).
  Arms: 8-mm shunt TIPS

SUMMARY:
Portal hypertension is the most common complication in patients with end-stage liver cirrhosis. Portal hypertension-related complications, such as variceal bleeding, often lead to a poor prognosis. Transjugular intrahepatic portosystemic shunt (TIPS) is an effective treatment strategy for managing portal hypertension-related variceal bleeding. However, the appropriate diameter of the covered stent during the TIPS procedure remains a subject of debate. To date, there is a lack of strong evidence regarding the most suitable covered stent diameter.

In theory, a shunt with a larger diameter can result in better stent patency, but it can also lead to reduced liver function and a higher incidence of hepatic encephalopathy (HE) after the TIPS procedure. Therefore, the choice of covered stent diameter needs to consider the factors of shunt efficacy and postoperative liver function. At present, the diameters of TIPS-dedicated stents are typically either 8 or 10 mm. Whether stents with these two diameters can meet all the requirements of TIPS procedures is currently unknown. Different races, cirrhosis etiologies, and liver volumes may require different TIPS diameters. For example, in China, most cases of liver cirrhosis are caused by hepatitis B, resulting in the patient having a smaller liver volume. Therefore, in most Chinese studies, the diameters of TIPS stents are mainly 8 mm. Previous studies have shown that TIPS with an 8-mm covered stent has a shunt effect similar to that of a 10-mm covered stent; however, the incidence of postoperative HE is significantly reduced with an 8-mm stent (27% vs. 43%)14. Nevertheless, an 8-mm covered TIPS still has a high incidence of HE.

The residual liver volume is small for patients with severe atrophic cirrhosis of the liver, and whether this necessitates a covered TIPS with a smaller diameter requires further study. However, there is still no dedicated TIPS stent that is <8 mm in diameter. In this study, we propose an innovative strategy for the creation of a 6-mm shunt to determine if it can achieve a shunt effect similar to that of an 8-mm covered TIPS and reduce the incidence of HE in patients with severe atrophic liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as cirrhosis
2. Previous or present endoscopic diagnosis of esophageal and gastric varices bleeding.
3. Child -Pugh score C (≤13) or MELD≤18.
4. Enhanced image measurement of liver volume ≤1000cm3.
5. Have indications for TIPS treatment.
6. Researchers believe that patients have the ability to comply with the research plan.
7. Sign the informed consent form

Exclusion Criteria:

1. Malignant tumor (including hepatocellular carcinoma) or other diseases that will shorten the life span of patients.
2. Cavernous portal vein
3. Non-cirrhotic portal hypertension (Budd-Chiari syndrome, extrahepatic portal vein obstruction, idiopathic portal hypertension, etc.)
4. Spontaneous dominant hepatic encephalopathy 5 congestive heart failure or severe valvular heart failure

6. Uncontrollable systemic infection or inflammation 7. Severe pulmonary hypertension 8. Severe renal insufficiency (except hepatogenic renal insufficiency) 9. Rapidly progressing liver failure 10. Contrast agent allergy 11. History of liver transplantation or allogeneic organ transplantation 12. Have a history of TIPS or shunt operation. 13. Pregnancy or lactation 14. Poor compliance 15. Participate in another clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
The 1- year rates of rebleeding | From receiving TIPS to one year after the end of treatment
The 2- year rates of rebleeding | From receiving TIPS to two year after the end of treatment

SECONDARY OUTCOMES:
The 1- year stent patency rates | From receiving TIPS to 1 year after the end of treatment
  During the follow-up, there was no thrombosis in the stent and complications related to portal hypertension caused by stent occlusion.
The 2- year stent patency rates | From receiving TIPS to 2 year after the end of treatment
  During the follow-up, there was no thrombosis in the stent and complications related to portal hypertension caused by stent occlusion.
The 1-year cumulative incidences of overt HE | From receiving TIPS to 1 year after the end of treatment
  HE greater than or equal to 2
The 2-year cumulative incidences of overt HE | From receiving TIPS to 2 year after the end of treatment
  HE greater than or equal to 2

IPD SHARING:
Plan to Share IPD: Yes
Incidence of rebleeding in 1 year and 2 years, incidence of overt hepatic encephalopathy in 1 year and 2 years, stent failure, incidence of hepatic encephalopathy, liver function (C-P score, ABI score), and overall survival.
Supporting Information: Study Protocol, SAP, ICF, CSR